CLINICAL TRIAL: NCT01251783
Title: Double Blind, Randomized, Controlled Clinical Trial for Evaluate The Efficiency and Safety of a Fiber System From Agave, With Prebiotic Action, Metlin® and Metlos®, Incorporated to an Infant Formula for Term Newborn Babies
Brief Title: A Prebiotic Agave Derivated Metlin & Metlos in Infant Formula
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Pediatrics, Mexico (Other Government)
Collaborators: Nekutli S.A. de C.V. (Unknown)
Responsible Party: Pedro Gutierrez Castrellon, National Pediatric of Pediatrics, Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Metlin&MetlosChildren
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Term Babies
Keywords: term babies
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Infant Formula (Active Comparator): Infant Formula without lactobaillus or Metlin or Metlos
  Interventions: Dietary Supplement: Infant Formula
- Fully breast milk (Active Comparator): Group non randomized with fully breast milk
  Interventions: Dietary Supplement: Exclusively breast milk
- Metlin+Metlos+Lactobacillus GG (Experimental): Infant Formula added with Metlin+Metlos (6g/L) and Lactobacillus GG 0.3x107UFC
  Interventions: Dietary Supplement: Metlin+metlos+Lactobacillus GG
- Metlin+Lactobacillus GG (Active Comparator): Infant Formula added with Metlin (6g/L) + Lactobacillus GG 0.3x107 UFC
  Interventions: Dietary Supplement: Metlin + Lactobacillus GG
- Metlos+Lactobacillus GG (Active Comparator): Infant Formula added with Metlos (6g/L)+Lactobacillus GG 0.3x107UFC
  Interventions: Dietary Supplement: Metlos + lactobacillus GG
- Lactobacillus GG (Active Comparator): Infant Formula added with Lactobacillus GG 0.3x107UFC without Metlin or Metlos
  Interventions: Dietary Supplement: Lactobacillus GG

INTERVENTIONS:
Dietary Supplement: Infant Formula — Only Infant Formula without Lactobacillus, Metlin OR Metlos
  Arms: Infant Formula
Dietary Supplement: Exclusively breast milk — Children non randomized which mothers decided to feed them with exclusively breast milk
  Arms: Fully breast milk
Dietary Supplement: Metlin+metlos+Lactobacillus GG — A prebiotic Agave Derivated Metlin+Metlos (6g/L) + 0.3x107 UFC Lactobacillus GG
  Arms: Metlin+Metlos+Lactobacillus GG
Dietary Supplement: Metlin + Lactobacillus GG — A prebiotic Agave Derivated Metlin (6g/L) + 0.3x107 UFC Lactobacillus GG
  Arms: Metlin+Lactobacillus GG
Dietary Supplement: Metlos + lactobacillus GG — A prebiotic Agave Derivated Metlos (6g/L) + 0.3x107 UFC Lactobacillus GG
  Arms: Metlos+Lactobacillus GG
Dietary Supplement: Lactobacillus GG — An Infant Formula added with 0.3x107 UFC Lactobacillus GG with no Metlin or Metlos
  Arms: Lactobacillus GG

SUMMARY:
Objectives: To evaluate the safety; efficacy; bone mineral metabolism & immunity changes of the use of Metlin & Metlos added to the Infant Formula Study Design: Randomized, double blind, clinical, controlled trial, in 600 full-term infants of 15 ± 7 days randomized to recive formula with probiotics + Metlin + Metlos; formula with probiotics + Metlin; Formula with probiotics + Metlos; formula only with probiotics or formula without probiotics and prebiotics; having a totally breast feed group as control.). Outcomes variables were frequency of stools; bowel intolerance manifestations (abdominal distension, flatulency, regurgitations, vomiting); report of dermatological problems like eczema; changes on the intestinal microbiota; lipids profile (cholesterol, triglycerides, lipoproteins associated to cholesterol); anthropomorphic profile and somatic growth ( weight gain, stature, arm mean circumference, skin folds); bone mineral metabolism (high-speed bone ultrasonography); and changes in the immunity (changes in the concentrations of salivary IgA and the frequency of respiratory events suggestive of infection)]. Statistical analysis was made with STATA Ver. 11.0 for Mac. Safety and efficacy variables, were compared by Chi squared in the case of categorical variables or by ANOVA or Kruskall Wallis for the numeric variables. When convenient, a covariates adjustment was done by ANOVA or by multiple lineal regressions for continuous numerical outcomes or logistic regression for categoric outcomes. In all the hypothesis tests the p significant value of <0.05 were used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term babies (37 to 42 weeks of gestationl age)
* Age 15 ± 7 days at admission
* Birth weight > 2,490 g.
* Negative history of formula intolerance (only randomized babies)
* Signed Informed Consent

Exclusion Criteria:

* Clinical evidence of chronic cardiac, respiratory, gastrointestinal, hematological or metabolic disease.
* Maternal medical history of diabetes (gestational diabetes was acceptable if the infant's birth weight was at or below the percentile 95; or 4153 g or 9 lbs 3 oz for girls or 4340 g or 9 lbs 9 oz for boys
* Tuberculosis, immunologic deficiency, infection disease or perinatal infections known to cause adverse effects in the fetus
* Participation in other study
* Inability of the father/mother or legal tutor to reed or comprehend the informed consent and the symtoms report diary, or
* The infant was part of multiple labor (twins, triplets, etc.)

Ages: 15 Days to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety of Metlin & Metlos Aministration in Infant Formula | February 2010 to September 2010
  Safety of Metlin & Metlos administration in infant formula was measured by means of the frequency of stools output reported daily by the mother or the keeper (nurse) during the whole study and by the presence gastrointestinal manifestations of intolerance (abdominal distension, flatulency, regurgitations, vomiting), or by the report of eczema type dermatological problems.

SECONDARY OUTCOMES:
Efficacy of Administration of Metlin & Metlos in Infant Formula | February 2010 to September 2010
  Efficacy of Metlin & Metlos in Infant Formula was measured by means of the change on the intestinal micro flora; changes in the lipids profile (cholesterol, triglycerides, lipoproteins associated to cholesterol); changes in the anthropomorphic profile and somatic growth ( weight gain, stature, arm mean circumference, skin folds); bone mineral metabolism (bone ultrasonography); changes in the immunity (changes in the concentrations of salivary IgA) and reduction of respiratory events suggestive of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Lopez-Vealzquez, PhD, Study Director — National Insitute of Pediatrics, Mexico; Pedro Gutierrez-Castrellon, MD, MSc, DSc, Principal Investigator — National Institute of Pediatrics, Mexico
Locations (1):
- National Pediatric Institute, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Leach JD, Sobolik KD. High dietary intake of prebiotic inulin-type fructans in the prehistoric Chihuahuan Desert. Br J Nutr. 2010 Jun;103(11):1558-61. doi: 10.1017/S0007114510000966. Epub 2010 Apr 26. PMID 20416127
- [Background] Gomez E, Tuohy KM, Gibson GR, Klinder A, Costabile A. In vitro evaluation of the fermentation properties and potential prebiotic activity of Agave fructans. J Appl Microbiol. 2010 Jun;108(6):2114-21. doi: 10.1111/j.1365-2672.2009.04617.x. Epub 2009 Nov 4. PMID 19941629
- [Background] Lopez MG, Mancilla-Margalli NA, Mendoza-Diaz G. Molecular structures of fructans from Agave tequilana Weber var. azul. J Agric Food Chem. 2003 Dec 31;51(27):7835-40. doi: 10.1021/jf030383v. PMID 14690361
- [Background] Gruber C, van Stuijvenberg M, Mosca F, Moro G, Chirico G, Braegger CP, Riedler J, Boehm G, Wahn U; MIPS 1 Working Group. Reduced occurrence of early atopic dermatitis because of immunoactive prebiotics among low-atopy-risk infants. J Allergy Clin Immunol. 2010 Oct;126(4):791-7. doi: 10.1016/j.jaci.2010.07.022. Epub 2010 Sep 15. PMID 20832848
- [Background] Sazawal S, Dhingra U, Hiremath G, Sarkar A, Dhingra P, Dutta A, Verma P, Menon VP, Black RE. Prebiotic and probiotic fortified milk in prevention of morbidities among children: community-based, randomized, double-blind, controlled trial. PLoS One. 2010 Aug 13;5(8):e12164. doi: 10.1371/journal.pone.0012164. PMID 20730056
- [Result] Sabater-Molina M, Larque E, Torrella F, Zamora S. Dietary fructooligosaccharides and potential benefits on health. J Physiol Biochem. 2009 Sep;65(3):315-28. doi: 10.1007/BF03180584. PMID 20119826
- [Derived] Lopez-Velazquez G, Parra-Ortiz M, Mora Ide L, Garcia-Torres I, Enriquez-Flores S, Alcantara-Ortigoza MA, Angel AG, Velazquez-Aragon J, Ortiz-Hernandez R, Cruz-Rubio JM, Villa-Barragan P, Jimenez-Gutierrez C, Gutierrez-Castrellon P. Effects of Fructans from Mexican Agave in Newborns Fed with Infant Formula: A Randomized Controlled Trial. Nutrients. 2015 Oct 29;7(11):8939-51. doi: 10.3390/nu7115442. PMID 26529006